CLINICAL TRIAL: NCT01822938
Title: Follow-up of Patients' Physical Activity in Post-hospitalization by Implementation of Systems of Active Monitoring.
Brief Title: Follow-up of Patients' Physical Activity in Post-hospitalization
Acronym: TICAA'DOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: I12006 / TICAA'DOM
Record Dates: First submitted 2013-03-25; First posted 2013-04-04 (Estimated); Last update posted 2018-08-14 (Actual); Status verified 2015-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- effects of a incentive program for physical activity (Experimental): The aim of the study is the assessment of the effects of a incentive program for physical activity on people following/with stroke
  Interventions: Other: incentive program for physical activity
- control group (No Intervention): No intervention

INTERVENTIONS:
Other: incentive program for physical activity
  Arms: effects of a incentive program for physical activity

SUMMARY:
Physical exercise has been identified as a major item of many affecting many chronic diseases and stroke rehabilitation. It contributes to an improvement in the quality of life and to a decrease in the current treatment side-effects and mortality. Stroke in association with an inactive lifestyle lead to a decrease in physical capability and causes problems in daily activities. The physical capacity and the tolerance for exercise fall simultaneously leading to vicious circle of less and less mobility. Therefore, physical activity for the health is a valid and relevant way to improve the quality of life and to recover functional capacity. The aim of the study is the assessment of the effects of a incentive program for physical activity on people following/with stroke.

ELIGIBILITY:
Inclusion Criteria:

* Person having stroke (ischemic or hemorrhagic)
* Whatever the area of stroke
* Person supported by HEMIPASS (monitoring team and home support)
* Stroke less than 6 months
* Patient walking with or without technical or human assistance: FCC score

Exclusion Criteria:

* Disability limiting the gait before the stroke
* Age < 18 years
* Cognitive impairment limiting participation to the program
* Non signature of the consent
* cardiopulmonary pathology which forbid/banned effort

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
The distance on the 6 minute walking test (6MWT) | 6 minutes

SECONDARY OUTCOMES:
Quality of life | at 0 month, 6 months and 12 months
  EQ-5D

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Limoges, Limoges, France

REFERENCES:
- [Derived] Guediri A, Chaparro D, Borel B, Daviet JC, Compagnat M, Mandigout S. The effect of a home-based coaching program on heart rate variability in subacute stroke patients: a randomized controlled trial. Int J Rehabil Res. 2022 Sep 1;45(3):201-208. doi: 10.1097/MRR.0000000000000529. Epub 2022 May 2. PMID 35502452
- [Derived] Mandigout S, Chaparro D, Borel B, Kammoun B, Salle JY, Compagnat M, Daviet JC. Effect of individualized coaching at home on walking capacity in subacute stroke patients: A randomized controlled trial (Ticaa'dom). Ann Phys Rehabil Med. 2021 Jul;64(4):101453. doi: 10.1016/j.rehab.2020.11.001. Epub 2020 Nov 28. PMID 33197648
- [Derived] Chaparro D, Daviet JC, Borel B, Kammoun B, Salle JY, Tchalla A, Mandigout S. Home-based physical activity incentive and education program in subacute phase of stroke recovery (Ticaa'dom): study protocol for a randomized controlled trial. Trials. 2018 Jan 25;19(1):68. doi: 10.1186/s13063-017-2410-9. PMID 29370824